CLINICAL TRIAL: NCT03003416
Title: Efficacy of Ozurdex® in the Treatment of Diabetic Macular Edema (DME)
Acronym: Louvre 3
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: GMA-EAME-EYE-0440
Record Dates: First submitted 2016-12-22; First posted 2016-12-28 (Estimated); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- OZURDEX®: Patients prescribed dexamethasone intravitreal implant (OZURDEX®) in clinical practice for the treatment of Diabetic Macular Edema.
  Interventions: Drug: dexamethasone intravitreal implant

INTERVENTIONS:
Drug: dexamethasone intravitreal implant — Dexamethasone intravitreal implant (OZURDEX®) as prescribed in clinical practice.
  Other Names: OZURDEX®

SUMMARY:
This study will evaluate the efficacy of Ozurdex® as prescribed in clinical practice in France for the treatment of Diabetic Macular Edema (DME).

ELIGIBILITY:
Inclusion Criteria:

-Patient with Diabetic Macular Edema (DME) treated with Ozurdex® in clinical practice.

Exclusion Criteria:

-Patient not residing in metropolitan France.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with OZURDEX® in clinical practice.
Sampling Method: Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2017-10-19 (Actual); Primary Completion 2018-12-19 (Actual); Study Completion 2018-12-19 (Actual)

PRIMARY OUTCOMES:
Best Gain in Best Corrected Visual Acuity (BCVA) compared to Baseline Using the Early Treatment Diabetic Retinopathy Study (ETDRS) Scale | Baseline to Month 24

SECONDARY OUTCOMES:
Time to Achieve Maximum Gain in BCVA | 24 Months
Change from Baseline in BCVA | Baseline, Week 6, Months 6, 12, 18 and 24
Percentage of Participants with a Gain (Improvement) in BCVA of at Least 10 Letters from Baseline | Baseline, Week 6, Month 6, 12, 18 and 24
Percentage of Participants with a Gain (Improvement) in BCVA of at Least 15 Letters from Baseline | Baseline, Week 6, Month 6, 12, 18 and 24
Change from Baseline in Retinal Thickness | Baseline, Month 24
Percentage of Participants with a 20% Reduction in Retinal Thickness compared to Baseline | Baseline, Month 24
Percentage of Participants with Disappearance of DME defined by Disappearance of Cyst or Obtaining a Normal Retinal Thickness | Month 24
Percentage of Participants Categorized by Demographic Characteristics Treated or Not Treated with Ozurdex® | Day 1
Percentage of Physicians Categorized by Age, Sex, Type of Practice, Number of Yearly Injections | Day 1
Percentage of Participants Categorized by Characteristics of Disease (DME or Diabetes) | Day 1
Percentage of Participants Categorized by Treatment Methods at Inclusion (Therapeutic Decision for inclusion or Reason for Non-Treatment) | Day 1
Percentage of Participants Categorized by Conditions when Placed on Treatment (Patient Characteristics, Glycosylated Hemoglobin (HbA1c) Level Control, Blood Pressure Control, Prior Treatments, Prior Treatment Failure) | Day 1
Percentage of Participants Categorized by Conditions when Use of Ozurdex® (Number of Injections, Number of Follow-up Visits, Criteria for Retreatment and Discontinuation of Treatment) | 24 Months
Percentage of Participants with at Least 1 Adverse Event (AE) based on intensity, relationship with the treatment and severity | 24 Months
Percentage of Participants by Intra-ocular Pressure (IOP) Categories (≥25 and ≥35 mmHg) | 24 Months
Number of Participants with Intra-ocular Pressure (IOP) Changes >10 mmHg from Baseline | 24 Months
Percentage of Participants Treated with a Hypotonic Agent, Laser, Filtration Surgery | 24 Months
Number of Participants with Incident Cataracts | 24 Months
Number of Participants with Cataract Surgeries Related to Treatment or Injection | 24 Months
Percentage of Participants with Serious Adverse Events | 24 Months
Percentage of Participants with Death | 24 Months

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Mesnard, Study Director — Allergan
Locations (25):
- France (25):
  - Centre MGM, Aix-en-Provence
  - Ballanger, Aulnay-sous-Bois
  - CH BLOIS, Blois
  - CH Avicennes Bobigny, Bobigny
  - Centre Rétine Gallien à Bordeaux, Bordeaux
  - CHU Bordeaux, Bordeaux
  - CHU Brest, Brest
  - CHI Créteil, Créteil
  - CH SCORFF - Lorient, Lorient
  - Hopital De La Croix Rousse, Lyon
  - Clinique Monticelli, Marseille
  - Hopital de la Timone, Marseille
  - CHR Annecy, Metz-Tessy
  - CHU Pasteur 2, Nice
  - Chno 1520, Paris
  - Hopital Saint Joseph, Paris
  - Fondation Rothschild, Paris
  - Lariboisiere, Paris
  - COCHIN, Paris
  - Hopital Poissy, Poissy
  - Hôpital de La Milétrie Poitiers, Poitiers
  - Hopital Saint Germain en Laye, Saint-Germain-en-Laye
  - Centre OPHTA.Kervision, Saint-Herblain
  - Maison Rouge, Strasbourg
  - Chu Toulouse, Toulouse

REFERENCES:
- [Derived] Kodjikian L, Delcourt C, Creuzot-Garcher C, Massin P, Conrath J, Velard ME, Lassalle T, Pinchinat S, Dupont-Benjamin L. Prospective, Observational, Multicenter, Real-World Study of the Efficacy, Safety, and Pattern of Use of the Dexamethasone Intravitreal Implant in Diabetic Macular Edema in France: Short-Term Outcomes of LOUVRE 3. Ophthalmol Ther. 2023 Jun;12(3):1671-1692. doi: 10.1007/s40123-023-00662-8. Epub 2023 Mar 26. PMID 36967448
- See also: More Information — http://www.allerganclinicaltrials.com